CLINICAL TRIAL: NCT02572141
Title: A Phase III Study to Evaluate the 3-year Disease-free Survival in Patients with Locally Advanced Colon Cancer Receiving Either Perioperative or Postoperative Chemotherapy with FOLFOX or CAPOX Regimens
Brief Title: FOLFOX or CAPOX Perioperative Chemotherapy Versus Postoperative Chemotherapy for Locally Advanced Colon Cancer (OPTICAL)
Acronym: OPTICAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Associate professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU10; C01 (Other: CSWOG)
Record Dates: First submitted 2015-10-01; First posted 2015-10-08 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Fluorouracil; Capecitabine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perioperative chemotherapy (Experimental): Perioperative chemotherapy with mFOLFOX6 or CAPOX regimens
  Interventions: Drug: Perioperative chemotherapy with mFOLFOX6 or CAPOX regimens
- Postoperative chemotherapy (Active Comparator): Postoperative chemotherapy with mFOLFOX6 or CAPOX regimens
  Interventions: Drug: Postoperative chemotherapy with mFOLFOX6 or CAPOX regimens

INTERVENTIONS:
Drug: Perioperative chemotherapy with mFOLFOX6 or CAPOX regimens — mFOLFOX6 (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-Fluorouracil 400 mg/m2 and IV infusional 5-Fluorouracil 2400 mg/m2 over 46h every 14 days) for 6 cycles followed by colectomy (3 to 5 weeks after) followed by mFOLFOX6 (6 cycles); CAPOX (IV oxaliplatin given over 120 min at a dose of 130 mg/m2 on day 1, oral capecitabine 1000 mg/m2 twice daily on days 1 through 14 every 21 days) for 4 cycles followed by colectomy (3 to 5 weeks after) followed by CAPOX (4 cycles).
  Other Names: Oxaliplatin; 5-Fluorouracil; Capecitabine; Leucovorin
  Arms: Perioperative chemotherapy
Drug: Postoperative chemotherapy with mFOLFOX6 or CAPOX regimens — Colectomy (maximum 4 weeks after randomization) followed by mFOLFOX6 (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-Fluorouracil 400 mg/m2 and IV infusional 5-Fluorouracil 2400 mg/m2 over 46h every 14 days) for 12 cycles; Colectomy (maximum 4 weeks after randomization) followed by CAPOX (IV oxaliplatin given over 120 min at a dose of 130 mg/m2 on day 1, oral capecitabine 1000 mg/m2 twice daily on days 1 through 14 every 21 days) for 8 cycles
  Other Names: Oxaliplatin; 5-Fluorouracil; Capecitabine; Leucovorin
  Arms: Postoperative chemotherapy

SUMMARY:
BACKGROUND:

In patients with high risk stage II and stage III colon cancer (CC), curative surgery followed by adjuvant chemotherapy with FOLFOX or CAPOX regimens has become a standard treatment. However, 20 to 30 % of these patients will develop distant metastasis, which ultimately result in death. Perioperative chemotherapy is a promising strategy with potential benefits that could be more effective at eradicating micrometastases. Moreover, shrinking tumor before surgery not only facilitate removal of all the tumor by the surgeon but also reduce tumor cell spreading during the procedure. With recent advances in radiology, preoperative computed tomography is a robust method for measuring the depth of tumor invasion and identifying the CC patients with poor prognosis, who may benefit from perioperative chemotherapy. The investigators conducted the present randomized study to explore whether perioperative chemotherapy with FOLFOX or CAPOX regimens compared with postoperative chemotherapy could improve disease-free survival in patients with radiologically staged, locally advanced, but resectable colon cancer.

OBJECTIVE:

The primary objective of this study is to evaluate the efficacy of perioperative chemotherapy with FOLFOX or CAPOX regimens compared to postoperative chemotherapy in patients with locally advanced colon cancer. Secondary objectives are efficacy in terms of R0 resection rate, overall survival (OS), relapse-free survival (RFS), down-staging of primary tumors, and tolerability of perioperative therapy and postoperative complications.

DETAILED DESCRIPTION:
OVERVIEW OF TRIAL DESIGN:

This trial is a a two-arm, multicenter, open labelled, prospective, randomized phase III studies. Eligible patients with locally advanced (T4 or T3 with extramural depth≧5 mm) colon cancer patients will be randomly assigned, in a 1:1 ratio, to receive either perioperative or postoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Histological or cytological documentation of adenocarcinoma of the colon (≥ 15 cm from the anal verge).
3. Determined preoperatively by either spiral or multidetector CT: high risk T3 (tumor disruption of muscle wall and extension into pericolic fat with more than 5 mm protrusion into adjacent mesenteric fat) or T4 (tumor penetrates to the surface of the visceral peritoneum or directly invades or is adherent to adjacent organs or structures).
4. Male or female subjects > 18 years < 70 of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. CT or MRI scans (done within 30 days of registration) of the chest, abdomen and pelvis all without clear evidence of distant metastatic (M1) disease.
7. Non complicated primary tumor (obstruction, perforation, bleeding).
8. No previous any systemic anticancer therapy for colon cancer disease.
9. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.
2. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
3. Heart failure grade III/IV (NYHA-classification).
4. Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
5. Subjects with known allergy to the study drugs or to any of its excipients.
6. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
7. Breast- feeding or pregnant women
8. Lack of effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years
  Defined as the time from randomization to relapse or death, whichever occurred first.

SECONDARY OUTCOMES:
Curative resection rate | 2 years
  Curative resection defined as complete tumor resection with all margins being negative.
Overall survival (OS) | 5 years
  Defined as the time from randomization to death from any cause.
Relapse-free survival (RFS) | 5 years
  Defined as the time from randomization to relapse.
Down-staging of primary tumors | 2 years
  Down-staging of the resected tumour as measured by histopathological tumour diameter and stage according to the TNM staging system of AJCC (7th version).
Toxicity assessed using the NCI common toxicity criteria, version 4.0. | 2 years
  The grade of toxicity will be assessed using the NCI common toxicity criteria, version 4.0.
Postoperative complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hu H, Zhang J, Li Y, Wang X, Wang Z, Wang H, Kang L, Liu P, Lan P, Wu X, Zhen Y, Pei H, Huang Z, Zhang H, Chen W, Zeng Y, Lai J, Wei H, Huang X, Chen J, Chen J, Tao K, Xu Q, Peng X, Liang J, Cai G, Ding K, Ding Z, Hu M, Zhang W, Tang B, Hong C, Cao J, Huang Z, Cao W, Li F, Wang X, Wang C, Huang Y, Zhao Y, Cai Y, Ling J, Xie X, Wu Z, Shi L, Ling L, Liu H, Wang J, Huang M, Deng Y; OPTICAL study group. Neoadjuvant Chemotherapy With Oxaliplatin and Fluoropyrimidine Versus Upfront Surgery for Locally Advanced Colon Cancer: The Randomized, Phase III OPTICAL Trial. J Clin Oncol. 2024 Sep 1;42(25):2978-2988. doi: 10.1200/JCO.23.01889. Epub 2024 Apr 2. PMID 38564700